CLINICAL TRIAL: NCT01983098
Title: Analysis of Circulating Tumor DNA to Monitor Metastatic Colorectal Cancer Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI-CRC-DNAc
Record Dates: First submitted 2013-10-28; First posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-10

CONDITIONS: To Compare the Monitoring of Circulating Tumor DNA With the Efficacy of Chemotherapy Evaluated by Computer Tomography Scan.
Keywords: Colorectal cancer; Metastatic; Circulating tumor DNA; Biomaker
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples were collected from patients treated for colorectal cancer. Blood samples were collected in EDTA tubes every two weeks before each cycles of chemotherapy. Blood samples were processed within 2 hour after collection and were centrifuged to separate the plasma from the peripheral-blood cells.
Oversight: Data Monitoring Committee: No

SUMMARY:
Colorectal cancer (CRC) is the third of the most common cancers and the second leading cause of cancer death in western countries. CRC is diagnosed at metastatic stage in approximately 35% of cases, while about 20% to 50% of patients diagnosed at earlier stage (stage II and III) will develop distant metastasis subsequently. Treatment efficacy is usually evaluated by computer tomography (CT) scan with RECIST criteria and dosage of carcinoembryonic antigen (CEA) and carbohydrate antigen (CA) 19-9, which were performed every two weeks during the chemotherapy. The management of treatment for metastatic CRC need the development of early biomarkers to evaluate the efficacy in order to avoid unnecessary toxicity in case of early chemotherapy resistance. In this prospective study, the investigators will compare the monitoring of circulating tumor DNA with the results of CT scan according the RECIST criteria and the blood level of CEA and CA 19-9. The investigators carried out a microfluidic digital polymerase-chain-reaction (PCR) assay to measure the specific somatic genomic alterations in plasma to identify the circulating tumor DNA.

DETAILED DESCRIPTION:
Description Colorectal cancer (CRC) is a real public health problem in the world. In Western countries, CRC is the third of the most common cancers and the second leading cause of cancer death. The prognosis of CRC is closely associated with the tumor stage at diagnosis. Despite widespread screening program, the CRC is diagnosed at metastatic stage in approximately 35% of cases, while about 20% to 50% of patients diagnosed at earlier stage (stage II and III) will develop distant metastasis subsequently. For these patients with metastatic CRC, improved surgical techniques, advances in cytotoxic chemotherapy regimens (fluoropyrimidin, oxaliplatin and irinotecan) and the progress of targeted therapies (antiangiogenic and anti-EGFR therapies) have increased survival and improve the quality of life. These patients are usually treated every 2 weeks with these chemotherapy regimens and the tumor response are evaluated every 2 months by computed tomography (CT) scan using the RECIST criteria (Therasse P, J Natl Cancer Inst 92:205-216, 2000). These morphological criteria determine several tumor response: complete remission (CR) is the disappearance of all lesions, partial response (PR) is the reduction of at least 30 % of the sum of the largest diameters of all lesions targets, progression disease (PD) is increased by at least 20 % of the sum of the largest diameters of target lesions or appearance of new lesions, and stable disease (SD) corresponds to the lower decrease in 30% or higher than 20 % of the sum of target lesions (P Therasse, J Natl Cancer Inst 92:205-216, 2000). Treatment should be changed in case of PD, while is usually continued in case of objective tumor response or control disease. Moreover, carcinoembryonic antigen (CEA) and carbohydrate antigen (CA) 19-9 are serum biomarkers that are clinically useful to evaluate efficacy of treatment in some patients with metastatic CRC but have a sensitivity of only 50 to 70%. Therefore, in case of early tumor resistance to treatment, PD will be objectified as CT scan only after 2 months of treatment, exposing the patient to unnecessary toxicity that could be sometimes severe. Early biomarkers of tumor response are needed for better management of treatment for patients with metastatic CRC.

CRC is characterized by highly specific genetic alterations. Some molecular alterations may be predictive (tailoring the protocols of chemotherapy) or prognostic (evaluating the severity of the disease) biomarkers useful in the therapeutic management of these patients. For example, KRAS tumor mutation was associated with a lack of response to anti-EGFR targeted therapies (Lievre A, J Clin Oncol 2008, 26:374-9; Lievre A, Cancer Res 2006,66:3992-5), while BRAF mutation are prognostic (Van Cutsem E, J Clin Oncol 2011, 29:2011-19). Specific genetic alterations in the tumor can also be detected from the circulating tumor DNA of patients with CRC (Lecomte T, Int J Cancer 2002, 100:543-8). Indeed, circulating DNA fragments carrying tumor specific sequence alterations (circulating tumor DNA) are found in the fraction of blood, representing a variable and generally small fraction of the total circulating DNA. Recently, a study showed that circulating tumor DNA was an informative, inherently specific, and highly sensitive biomarker of monitoring for metastatic breast cancer treatment (N Engl J Med. 2013;368:1199-209). However, to our knowledge, analysis of circulating tumor DNA to monitor metastatic CRC was not performed yet. The aim of our study is to determine a biomarker evaluating precociously the response to chemotherapy by the monitoring of the circulating tumor DNA.

Patients and Methods Results of CT imaging, levels of CEA and CA 19-9, and serial whole-blood samples were collected prospectively from patients undergoing therapy for metastatic CRC. DNA extracted from archival tumor tissue samples was analysed to identify somatic genomic alterations (KRAS, NRAS, BRAF, TP53, PI3KCA, APC, SMAD4 …). Blood samples were collected in EDTA tubes every two weeks before each cycles of chemotherapy. Blood samples were processed within 2 hour after collection and were centrifuged to separate the plasma from the peripheral-blood cells. DNA was extracted from plasma. To measure the DNA carrying specific somatic genomic alterations in plasma, the investigators carried out a microfluidic digital polymerase-chain-reaction (PCR) assay (Taly V, Clin Chem 2013).

The investigators will compare the monitoring of circulating tumor DNA with the results of CT scan according the RECIST criteria and the blood level of CEA and CA 19-9.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 ans,
* histologically proven metastatic colorectal adenocarcinoma,
* at least one measurable lesion (RECIST criteria),
* strating a new line of chemotherapy including fluoropyrimidin and/or oxaliplatin and/or irinotecan with or without targeted therapy(EGFR-targeted therapy or antiangiogenic), and written informed consent.

Exclusion Criteria:

* Patient unable to read or understand and sign the information sheet and consent form
* Patient not insured under the social security

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 18 ans treated in our center (European Georges Pompidou Hospital) by chemotherapy for metastatic colorectal cancer
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
To compare the monitoring of circulating tumor DNA with the results of computer tomography scan according the RECIST criteria | From first biomarker date to first clinical event
To compare the monitoring of circulating tumor DNA with the response tumor evaluated by RECIST criteria on computer tomography scan | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Aziz ZAANAN, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - HEGP, Paris
  - Hopital Européen Georges Pompidou, Paris

REFERENCES:
- [Derived] Unseld M, Belic J, Pierer K, Zhou Q, Moser T, Bauer R, Piringer G, Gerger A, Siebenhuner A, Speicher M, Heitzer E, Prager GW. A higher ctDNA fraction decreases survival in regorafenib-treated metastatic colorectal cancer patients. Results from the regorafenib's liquid biopsy translational biomarker phase II pilot study. Int J Cancer. 2021 Mar 15;148(6):1452-1461. doi: 10.1002/ijc.33303. Epub 2020 Oct 16. PMID 32949150